CLINICAL TRIAL: NCT00635492
Title: CHOICE: CHanges to Treatment and Outcomes in Patients With Type 2 Diabetes Initiating InjeCtablE Therapy - A European Observational Study of Patients With Type 2 Diabetes Initiating Injectable Therapy to Determine Time to Treatment Change, Factors Associated With Treatment Changes and Outcomes Over 24 Months
Brief Title: CHOICE: CHanges to Treatment and Outcomes in Patients With Type 2 Diabetes Initiating InjeCtablE Therapy
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: H8O-EW-B005
Record Dates: First submitted 2008-02-20; First posted 2008-03-13 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; insulin; exenatide; Byetta; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Exenatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: exenatide
  Interventions: Drug: exenatide
- 2: insulin
  Interventions: Drug: any human insulin or analog insulin(s) given in any regimen by subcutaneous injection

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day
  Other Names: Byetta
  Groups: 1
Drug: any human insulin or analog insulin(s) given in any regimen by subcutaneous injection
  Groups: 2

SUMMARY:
Patients initiating injectable therapy for type 2 diabetes (insulin or exenatide) in usual clinical practice will be enrolled and followed up for two years in order to describe actual practice with regards to the time on initial treatment regime, whether treatment regimens are being modified, what treatment modifications are made, and clinical and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* are aged 18 or above
* diagnosed with type 2 diabetes
* have had a treatment decision made within the normal course of care to initiate either insulin or exenatide for the treatment of type 2 diabetes
* have not previously been treated with either insulin or exenatide
* are not simultaneously participating in another study which includes an investigational drug or procedure at study entry
* have been fully informed and given their written consent for use of their data
* have sufficient understanding of the primary language of their country such that they will be able to complete the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients aged 18 or above, with type 2 diabetes starting any of the available initial injectable treatment options (any insulin, or exenatide BID) for the treatment of type 2 diabetes as part of routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 2515 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (96):
- Denmark (2):
  - Research Site, Amager
  - Research Site, Rønne
- Research Site, Toul, France
- Germany (76):
  - Research Site, Alsfeld
  - Research, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Aßlar
  - Research Site, Bad Aibling
  - Research Site, Bad Homburg
  - Research Site, Bad Mergentheim
  - Research Site, Bergheim
  - Research Site, Berlin
  - Research, Birkenfeld
  - Research Site, Bosenheim
  - Research Site, Bruchsal
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Eberswalde
  - Research Site, Eilenburg
  - Research Site, Eisenach
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Gebhardshain
  - Research Site, Gersfeld
  - Research Site, Giessen
  - Research Site, Gifhorn
  - Research Site, Grassau
  - Research Site, Groß-Gerau
  - Research Site, Hadmersleben
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hammelburg
  - Research Site, Hennigsdorf
  - Research Site, Hohenmölsen
  - Research Site, Ismaning
  - Research Site, Köthen
  - Research Site, Kutenholz
  - Research Site, Langen
  - Research Site, Langenfeld
  - Research Site, Leipzig
  - Research Site, Lichtenfels
  - Research Site, Ludwigsburg
  - Research Site, Lüneburg
  - Research Site, Marburg
  - Research Site, Mayen
  - Research Site, Meissen
  - Research Site, Minden
  - Research Site, Mönchengladbach
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nassau
  - Research Site, Netphen
  - Research Site, Oberhausen
  - Research Site, Pirmasens
  - Research Site, Recklinghausen
  - Research Site, Rehburg-Loccum
  - Research Site, Reichenbach
  - Research Site, Riesa
  - Research Site, Saarbrücken
  - Research Site, Saarlouis
  - Research Site, Schkeuditz
  - Research Site, Schönwalde
  - Research Site, Schweinfurt
  - Research Site, Seligenstadt
  - Research Site, Siegen
  - Research Site, Stockach
  - Research Site, Thale
  - Research Site, Ueckermünde
  - Research Site, Übach-Palenberg
  - Research Site, Villingen-Schwenningen
  - Research Site, Völklingen
  - Research Site, Warburg
  - Research Site, Weißenberg
  - Research Site, Werl
  - Research Site, Westfalica
  - Research Site, Wilhelmshaven
  - Research Site, Wurzen
- Greece (4):
  - Research Site, Kozani
  - Research Site, N. Efkarpia
  - Research Site, Thessaloniki
  - Research Site, Véroia
- Sweden (13):
  - Research Site, Angered
  - Research Site, Ängelholm
  - Research Site, Dalby
  - Research Site, Falun
  - Research Site, Gothenburg
  - Research Site, Limhamn
  - Research Site, Luleå
  - Research Site, Malmo
  - Research Site, Skivarp
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Vadstena
  - Research Site, Västervik

REFERENCES:
- [Derived] Schultheis P, Montoya MN, Zhao Q, Archer J, Madden T, Peipert JF. Contraception and ectopic pregnancy risk: a prospective observational analysis. Am J Obstet Gynecol. 2021 Feb;224(2):228-229. doi: 10.1016/j.ajog.2020.10.013. Epub 2020 Oct 10. No abstract available. PMID 33049248
- [Derived] Reaney M, Mathieu C, Ostenson CG, Matthaei S, Krarup T, Kiljanski J, Salaun-Martin C, Sapin H, Theodorakis M, Guerci B. Patient-reported outcomes among patients using exenatide twice daily or insulin in clinical practice in six European countries: the CHOICE prospective observational study. Health Qual Life Outcomes. 2013 Dec 26;11:217. doi: 10.1186/1477-7525-11-217. PMID 24369764
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study was conducted at 322 study centers in 6 countries (Belgium, Denmark, France, Germany, Greece, Sweden).
  Date of first patient enrolled: 25 January 2008 Date of last patient completed: 01 December 2011
Pre-assignment Details: 2515 patients enrolled. 2388 patients in final analysis (22 not in either cohort), excluded: 92 had no investigator signature on summary page, 11 had no treatment start date, 2 had issues with their informed consent to release their data.
Groups:
- Exenatide BID: Daily dose ranging from 5-20 mcg
- Insulin: Insulin at a dose selected by the health care provided (HCP) and patient
Period: Overall Study
Arm/Group | Exenatide BID | Insulin
Started | 1114 (This population consists of the analysis population.) | 1274 (This population consists of the analysis population.)
Completed | 835 (This population consists of patients that completed the 24 month study.) | 992 (This population consists of patients that completed the 24 month study.)
Not Completed | 279 | 282
Not completed — Death | 12 | 40
Not completed — Lost to Follow-up | 151 | 172
Not completed — Physician Decision | 32 | 22
Not completed — Sponsor decision | 2 | 3
Not completed — Withdrawal by Subject | 82 | 45

BASELINE CHARACTERISTICS:
Population: Analysis population description: all patients who provided consent to release information and who fulfill the study entry criteria were included in the analyses. Patients were assigned to the exenatide BID or insulin cohort based on their initial injectable treatment started at baseline.
Groups:
- Exenatide BID: Daily dose ranging from 5-20 ug
- Insulin: Insulin at a dose selected by the HCP and patient
- Total: Total of all reporting groups
Arm/Group | Exenatide BID | Insulin | Total
Number analyzed (Participants) | 1114 | 1274 | 2388
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.1) | 63.7 (10.9) | 61.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 516 | 541 | 1057
  Male | 598 | 733 | 1331
Region of Enrollment [Number; unit: participants]
  France | 168 | 84 | 252
  Greece | 319 | 488 | 807
  Denmark | 43 | 16 | 59
  Germany | 384 | 438 | 822
  Sweden | 84 | 85 | 169
  Belgium | 116 | 163 | 279
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.4 (1.4) | 9.2 (1.9) | 8.8 (1.7)
Body Weight [Mean (Standard Deviation); unit: kg] | 101.2 (21.8) | 84.2 (17.6) | 92.1 (21.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 35.3 (6.6) | 29.7 (5.4) | 32.3 (6.6)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 8.2 (5.7) | 9.8 (7.3) | 9.1 (6.7)
Concomitant Oral Anti-Diabetic Medication [Number; unit: Number of Patients] — Number of patients on oral antidiabetic (OAD) medication at baseline. No differentiation possible if patients who did not report OADs actually took no OADs or just did not report them.
  Number of Patients
    No OAD | 50 | 154 | 204
    Single OAD | 383 | 476 | 859
    Combination of 2 OADs | 552 | 523 | 1075
    Combination of 3 OADs | 118 | 112 | 230
    Combination of 4 OADs | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Estimates of Probability to Remain on Initial Injectable Treatment at 12 and 24 Months.
Description: The primary objective of this study is to estimate the time spent on initial treatment regime before significant treatment change for patients with type 2 diabetes initiating therapy with either insulin or exenatide for the first time.
  Initial treatment regime is defined as the treatment regime prescribed when the patient is enrolled in the study.
  Significant treatment change for patients initiated on insulin or exenatide is defined as at least one of the following:
  Insulin:
  * Addition of a new medication for the treatment of type 2 diabetes
  * A change in the number of times insulin is administered per day
  * Discontinuation of any insulin initiated at baseline
  * Substitution of a human insulin for an analogue insulin or vice-versa.
  * Switching between brands of the same class/type of insulin is not included in the definition of significant treatment change.
  Exenatide:
  * Addition of a new medication for the treatment of type 2 diabetes
  * Discontinuation of exenatide.
Time Frame: Month 24
Population: All patients who provided consent to release information and who fulfil the study entry criteria were included in the analyses. Patients were assigned to the exenatide BID or insulin cohort based the injectable treatment started at baseline; analyses were conducted irrespective of later treatment changes.
Measure: Number (95% Confidence Interval); unit: probability (%)
Groups:
- Exenatide BID: daily dose ranging from 5-20mcg/day
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1113 | 1273
probability (%)
  Estimate at 24 months | 53.9 (123) [50.8 to 57.0] | 60.6 (123) [57.7 to 63.5]
  Estimate at 12 months | 67.8 [65.0 to 70.6] | 70.6 [68.0 to 73.1]

2. Secondary Outcome: Higher Body Mass Index (BMI) Associated With Treatment Choice at Baseline
Description: Higher BMI was one of the Factors evaluated for association with treatment choice at baseline. BMI was calculated as body weight in kilograms (kg) divided by height in meters (m) squared (kg/m^2). The mean BMI at baseline is provided below and the statistical analysis provides the 2 arms odds ratio for BMI=1 kg/m^2 higher. Participants were assigned to the exenatide BID or insulin cohort based the injectable treatment started at baseline; analyses were conducted irrespective of later treatment changes. Baseline was Visit T1 (prior to start of treatment).
Time Frame: Baseline
Population: All participants who provided consent to release information, fulfilled the study entry criteria, and had a start date provided were included in the analyses.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1177 | 1315
kg/m^2 | 35.3 (6.5) [1.13 to 1.19] | 29.7 (5.4)
Statistical Analysis 1: Comparison: Exenatide BID vs Insulin; Body Mass Index (BMI) - 1kg/m² higher; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [1.13 to 1.19]

3. Secondary Outcome: Higher Hemoglobin A1c (HbA1) Associated With Treatment Choice at Baseline
Description: Higher HbA1c was one of the Factors evaluated for association with treatment choice at baseline.HbA1c was reported in percent of hemoglobin. The mean HbA1c at baseline is provided below and the statistical analysis provides the 2 arms odds ratio for HbA1c=1% higher.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent of hemoglobin
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1177 | 1315
percent of hemoglobin | 8.4 (1.4) | 9.2 (1.9)
Statistical Analysis 1: Comparison: Exenatide BID vs Insulin; Most recent HbA1c at baseline - 1% higher; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.69 to 0.86]

4. Secondary Outcome: Older Age Associated With Treatment Choice at Baseline
Description: Older age (1 year older) was one of the Factors evaluated for association with treatment choice at baseline. The mean age at baseline is provided below and the statistical analysis provides the 2 arms odds ratio for age 1 year older. Participants were assigned to the exenatide BID or insulin cohort based the injectable treatment started at baseline; analyses were conducted irrespective of later treatment changes. Baseline was Visit T1 (prior to start of treatment).
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1114 | 1274
years | 58.1 (10.1) | 63.7 (10.9)
Statistical Analysis 1: Comparison: Exenatide BID vs Insulin; Age - 1 year older; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.95 to 0.97]

5. Secondary Outcome: Disinhibited Eating Associated With Treatment Choice at Baseline
Description: Diabetes Health Profile (DHP-18) - consists of 18 items across 3 domains (psychological distress, barriers to activity, and disinhibited eating), with each item standardized score rated from 0-100; 0=no dysfunction, higher numbers=greater dysfunction. The subscale of disinhibited eating was one of the Factors evaluated for association with treatment choice at baseline. The number of participants with disinhibited eating at baseline is provided below and the statistical analysis provides the 2 arms odds ratio for disinhibited eating. Participants were assigned to the exenatide BID or insulin cohort based the injectable treatment started at baseline; analyses were conducted irrespective of later treatment changes. Baseline was Visit T1 (prior to start of treatment).
Time Frame: Baseline
Population: All participants who provided consent to release information, fulfilled the study entry criteria, provided the specific data (DHP-18 subscale on disinhibited eating) and had a start date provided were included in the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 386 | 446
units on a scale | 43.52 (20.99) | 34.38 (20.33)
Statistical Analysis 1: Comparison: Exenatide BID vs Insulin; Diabetes Health Profile - 18 (DHP-18) subscale disinhibited eating - Yes vs. No; Test type: Superiority or Other; p = 0.0083, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [1.01 to 1.10]

6. Secondary Outcome: Higher Random Glucose Associated With Treatment Choice at Baseline
Description: Random Glucose 1 millimole per liter (mmol/L) higher was one of the Factors evaluated for association with treatment choice at baseline. Random glucose is a glucose within the last 6 months prior to baseline. The mean is provided below and the statistical analysis provides the 2 arms odds ratio for the glucose 1 mmol/L higher. Participants were assigned to the exenatide BID or insulin cohort based the injectable treatment started at baseline; analyses were conducted irrespective of later treatment changes. Baseline was Visit T1 (prior to start of treatment).
Time Frame: 6 months prior to Baseline
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1177 | 1315
mmol/L | 10.37 (3.13) | 12.13 (4.36)
Statistical Analysis 1: Comparison: Exenatide BID vs Insulin; Random blood glucose - 1 mmol/L higher; Test type: Superiority or Other; p = 0.0141, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.90 to 0.99]

7. Secondary Outcome: Frequent Blood Glucose Self Monitoring Associated With Treatment Choice at Baseline
Description: Frequent glucose self-testing (1 test/week more) was one of the Factors evaluated for association with treatment choice at baseline. The mean number of self monitoring blood glucose tests per week over the last 4 weeks prior to baseline was determined at baseline and is provided below. The statistical analysis provides the 2 arms odds ratio. Participants were assigned to the exenatide BID or insulin cohort based the injectable treatment started at baseline; analyses were conducted irrespective of later treatment changes. Baseline was Visit T1 (prior to start of treatment).
Time Frame: 4 weeks prior to Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tests/week
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 928 | 1050
tests/week | 9.28 (7.98) | 9.91 (8.58)
Statistical Analysis 1: Comparison: Exenatide BID vs Insulin; Blood glucose self-monitoring - 1 test/week more; Test type: Superiority or Other; p = 0.0107, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.96 to 0.99]

8. Secondary Outcome: Diet and Exercise Advice in Diabetes Management Associated With Treatment Choice at Baseline
Description: Receipt of diet and exercise advice was one of the Factors evaluated for association with treatment choice at baseline. The number of participants who checked yes or no during the baseline visit for prior receipt of diet/exercise advice in his/her Diabetes management is provided below and the statistical analysis provides the 2 arms odds ratio. Participants were assigned to the exenatide BID or insulin cohort based the injectable treatment started at baseline; analyses were conducted irrespective of later treatment changes. Baseline was Visit T1 (prior to start of treatment).
Time Frame: Baseline
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1177 | 1315
participants
  Missing | 12 | 1
  No | 131 | 237
  Yes | 910 | 905
  Unknown | 124 | 172
Statistical Analysis 1: Comparison: Exenatide BID vs Insulin; Receipt of diet/exercise advice - Yes vs. No; Test type: Superiority or Other; p = 0.0193, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.13 to 2.46]

9. Secondary Outcome: Higher Value of Low Density Lipoprotein Cholesterol Associated With Treatment Choice at Baseline
Description: Higher (1 mmol/L higher) LDL cholesterol was one of the Factors evaluated for association with treatment choice at baseline. The mean LDL cholesterol at baseline is provided below and the statistical analysis provides the 2 arms odds ratio for 1 mmol/L higher at baseline. Participants were assigned to the exenatide BID or insulin cohort based the injectable treatment started at baseline; analyses were conducted irrespective of later treatment changes. Baseline was Visit T1 (prior to start of treatment).
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1177 | 1315
mmol/L | 2.82 (1.09) | 3.00 (1.01)
Statistical Analysis 1: Comparison: Exenatide BID vs Insulin; LDL cholesterol - 1 mmol/L higher at baseline; Test type: Superiority or Other; p = 0.0138, Regression, Logistic; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.72 to 0.96]

10. Secondary Outcome: Changes in HbA1c From Baseline to Month 24
Description: Changes in HbA1c From Baseline to Month 24
Time Frame: Baseline, Month 24
Population: Patients were assigned to the exenatide BID or insulin cohort based on their initial injectable treatment started at baseline, and analyses were conducted irrespective of later treatment changes.
  All patients who provided consent to release information and who fulfilled study entry criteria were included in this analysis population.
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 795 | 924
percentage of total hemoglobin | -1.03 (1.48) | -1.71 (1.82)

11. Secondary Outcome: Percentage of Patients Achieving HbA1c Concentration <7.0% at Month 24
Description: Percentage of Patients Achieving HbA1c Concentration <7.0% at Month 24. Only patients with baseline HbA1c >= 7.0 % were included in this analysis
Time Frame: Month 24
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 959 | 1170
percentage of patients | 26.9 | 28.5

12. Secondary Outcome: Percentage of Patients Achieving HbA1c Concentration <6.5% at Month 24
Description: Percentage of Patients Achieving HbA1c Concentration <6.5% at Month 24. Note: Only patients with baseline HbA1c >=6.5% were included in this analysis.
Time Frame: Month 24
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1019 | 1208
percentage of patients | 12.5 | 10.7

13. Secondary Outcome: Changes in Weight From Baseline to Month 24
Description: Changes in Weight From Baseline to Month 24
Time Frame: Baseline, Month 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 810 | 945
kg | -3.22 (7.93) | 2.16 (6.24)

14. Secondary Outcome: Incidence of Gastro Intestinal Symptoms Between Baseline and 24 Months
Description: Incidence of Gastro Intestinal Symptoms between Baseline and 24 Months
Time Frame: Baseline to Month 24
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1114 | 1274
percentage of patients | 29.4 | 5.0

15. Secondary Outcome: Incidence of Hypoglycemia Between Baseline and 24 Months
Description: Incidence of Hypoglycemia between Baseline and 24 Months
Time Frame: Baseline to Month 24
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1114 | 1274
percentage of patients | 17.5 | 35.2

16. Secondary Outcome: Reasons for Discontinuation of Baseline Regimen
Description: Reasons for Discontinuation of Baseline Regimen
Time Frame: Baseline to Month 24
Population: as for outcome 10
Measure: Number; unit: number of patients
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 393 | 155
number of patients
  Inadequate response | 170 | 87
  Adverse event | 91 | 11
  Patient decision | 69 | 15
  Non compliance | 9 | 3
  Cannot afford medication | 4 | 1
  Other | 50 | 38

17. Secondary Outcome: Factors Associated With Treatment Change in Insulin Cohort
Description: Hazards ratios from Backward Cox Regression Model for time to significant treatment change in Insulin cohort
Time Frame: Baseline to Month 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: hazard ratio
Groups:
- Insulin Cohort: insulin at a dose selected by the HCP and patient
Arm/Group | Insulin Cohort
Number analyzed (Participants) | 1180
hazard ratio
  HbA1c (%) at baseline | 1.118 [1.062 to 1.177]
  DHP barriers to activity subscale at baseline | 0.960 [0.937 to 0.985]
  Gastrointestinal symptoms: yes vs. no at baseline | 2.532 [1.698 to 3.777]
  Insulin regimen: basal/bolus vs. long-acting only | 0.437 [0.303 to 0.630]
  Insulin regimen: mixtures vs. long-acting only | 0.676 [0.523 to 0.874]
  Insulin regimen: other vs. long-acting only | 0.549 [0.175 to 1.718]
  Insulin regimen: short-acting only vs. long-actin | 2.164 [1.681 to 2.785]
Statistical Analysis 1: Comparison: Insulin Cohort; HbA1c (%) at baseline; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 1.118, 95% CI 2-sided [1.062 to 1.177]
Statistical Analysis 2: Comparison: Insulin Cohort; DHP barriers to activity subscale at baseline; Test type: Superiority or Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 0.960, 95% CI 2-sided [0.937 to 0.985]
Statistical Analysis 3: Comparison: Insulin Cohort; Gastrointestinal symptoms: yes vs. no at baseline; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.532, 95% CI 2-sided [1.698 to 3.777]
Statistical Analysis 4: Comparison: Insulin Cohort; Insulin regimen: basal/bolus vs. long-acting only; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.437, 95% CI 2-sided [0.303 to 0.630]
Statistical Analysis 5: Comparison: Insulin Cohort; Insulin regimen: mixtures vs. long-acting only; Test type: Superiority or Other; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 0.676, 95% CI 2-sided [0.523 to 0.874]
Statistical Analysis 6: Comparison: Insulin Cohort; Insulin regimen: other vs. long-acting only; Test type: Superiority or Other; p = 0.303, Regression, Cox; Hazard Ratio (HR) = 0.549, 95% CI 2-sided [0.175 to 1.718]
Statistical Analysis 7: Comparison: Insulin Cohort; Insulin regimen: short-acting only vs. long-acting only; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.164, 95% CI 2-sided [1.681 to 2.785]

18. Secondary Outcome: Factors Associated With Treatment Change in Exenatide BID Cohort
Description: Hazards ratios from Backward Cox Regression Model for time to significant treatment change in Exenatide BID cohort. EQ-5D (Health Questionnaire Copyright @ Euro QoL Group 1998).
Time Frame: Baseline to Month 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Exenatide BID
Number analyzed (Participants) | 1019
hazard ratio
  Gastro intestinal symptoms: yes vs no at baseline | 1.463 [1.043 to 2.053]
  EQ-5D index value at baseline | 0.601 [0.432 to 0.834]
Statistical Analysis 1: Comparison: Exenatide BID; GI symptoms: yes vs. no at baseline; Test type: Superiority or Other; p = 0.028, Regression, Cox; Hazard Ratio (HR) = 1.463, 95% CI 2-sided [1.043 to 2.053]
Statistical Analysis 2: Comparison: Exenatide BID; EQ-5D index value at baseline; Test type: Superiority or Other; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.601, 95% CI 2-sided [0.432 to 0.834]

19. Secondary Outcome: Percentage of Patients Contacting Health Care Providers Between Baseline and 24 Months
Description: Percentage of Patients Contacting Health Care Providers Between Baseline and 24 Months
Time Frame: Baseline to Month 24
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1114 | 1274
percentage of patients
  Last 6 months prior to baseline | 94.4 | 94.1
  Baseline to 24 months | 90.4 | 92.3

20. Secondary Outcome: Number of Contacts With Health Care Providers Between Baseline and 24 Months
Description: Number of contacts with Health Care Providers Between Baseline and 24 Months
Time Frame: Baseline to Month 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: number of contacts
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1114 | 1274
number of contacts
  Last 6 months prior to baseline | 7.17 (6.92) | 7.64 (8.51)
  Baseline to 24 months | 19.00 (18.20) | 24.58 (32.75)

21. Secondary Outcome: Percentage of Patients Hospitalized Between Baseline and 24 Months
Description: Percentage of Patients Hospitalized Between Baseline and 24 Months
Time Frame: Baseline to Month 24
Population: as for outcome 10
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide BID | Insulin
Number analyzed (Participants) | 1114 | 1274
percentage of patients
  Last 6 months prior to baseline | 4.7 | 6.4
  Baseline to 24 months | 4.3 | 7.8

ADVERSE EVENTS:
Arm/Group | Exenatide BID | Insulin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
1. Serious adverse events (SAEs) and adverse events (AEs) were not collected as part of this observational study
2. Factors associated with treatment choice : this analysis was done on baseline lock( april 2009) where all others are from final lock.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.